CLINICAL TRIAL: NCT05584657
Title: A Prospective, Phase 3, Randomized, Multi-center, Double-blind Study of the Efficacy, Tolerability, and Safety of Oral Sulopenem Etzadroxil/Probenecid Versus Oral Amoxicillin/Clavulanate for Treatment of Uncomplicated Urinary Tract Infections (uUTI) in Adult Women
Brief Title: Oral Sulopenem Versus Amoxicillin/Clavulanate for Uncomplicated Urinary Tract Infection in Adult Women
Acronym: REASSURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Iterum Therapeutics, International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IT001-310
Expanded Access: NCT04682834 (No longer available)
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Urinary Tract Infections; Cystitis
MeSH Terms: conditions — Urinary Tract Infections; Cystitis | interventions — Probenecid; sulopenem; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sulopenem etzadroxil/probenecid (Experimental): Sulopenem etzadroxil/probenecid 500 mg/500 mg PO twice daily for 5 days
  Interventions: Drug: Sulopenem etzadroxil/probenecid
- Amoxicillin/clavulanate (Active Comparator): Amoxicillin/clavulanate PO twice daily for 5 days
  Interventions: Drug: Amoxicillin/clavulanate

INTERVENTIONS:
Drug: Sulopenem etzadroxil/probenecid — Oral sulopenem twice daily for 5 days
  Other Names: Oral sulopenem
  Arms: Sulopenem etzadroxil/probenecid
Drug: Amoxicillin/clavulanate — Oral Augmentin twice daily for 5 days
  Other Names: Augmentin
  Arms: Amoxicillin/clavulanate

SUMMARY:
Study 310 is a clinical study which compares the effectiveness of oral sulopenem versus oral amoxicillin/clavulanate for the treatment of adult women with uncomplicated urinary tract infection.

DETAILED DESCRIPTION:
IT001-310 is a Phase 3, randomized, multicenter, double-blind, double dummy, controlled study to compare oral sulopenem etzadroxil/probenecid (oral sulopenem) to oral amoxicillin/clavulanate for the treatment of adult female patients with uncomplicated urinary tract infection. Approximately 1966 adult women with uncomplicated urinary tract infection will be randomized in a 1:1 fashion to receive either oral sulopenem etzadroxil/probenecid or oral amoxicillin/clavulanate twice daily for 5 days. The primary outcome measure for efficacy evaluation will be the overall success (combined clinical and microbiologic success) on Day 12 (± 1 day)/Test of Cure (TOC).

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥18 years of age with ≥24 hours and ≤96 hours of urinary symptoms attributable to a UTI
* Two of the following signs and symptoms of uUTI: urinary frequency, urinary urgency, pain or burning on micturition, suprapubic pain.
* A mid-stream urine specimen with evidence of pyuria as defined by either a machine-read dipstick positive for leukocyte esterase OR at least 10 white blood cells per cubic millimeter on microscopic analysis of unspun urine OR white blood cell count ≥10 cells/high-powered field (HPF) in the sediment of a spun urine

Exclusion Criteria:

* Presence of signs and symptoms suggestive of acute pyelonephritis defined as: fever (temperature > 38° Celsius), chills, costovertebral angle tenderness, flank pain, nausea, and/or vomiting
* Receipt of antibacterial drug therapy potentially effective as treatment of uUTI within the prior 7 days
* Concurrent use of non-study treatments that would have a potential effect on outcome evaluations in patients with uUTI, including analgesics (e.g., non-steroidal anti-inflammatory drugs, aspirin, paracetamol etc.), phenazopyridine, and cranberry products.
* Any anatomical abnormality of the urinary tract, including surgically modified urinary tract anatomy, and obstructive uropathy due to nephrolithiasis, stricture, tumor, or fibrosis
* Ongoing urinary retention
* Neurogenic bladder
* Current resident of a long-term care facility
* Instrumentation of urinary tract in the previous 30 days
* An indwelling urinary catheter, ureteral stent or other foreign material in the urinary tract
* Any history of trauma to the pelvis or urinary tract
* Receiving hemodialysis, hemofiltration, peritoneal dialysis, or had a renal transplant
* History of allergy or hypersensitivity to carbapenems, β-lactams or probenecid, as formulated with their excipients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2229 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sailaja Puttagunta, MD, Study Director — Iterum Therapeutics
Locations (167):
- United States (167):
  - Medical Facility, Cullman, Alabama
  - Medical Facility, Saraland, Alabama
  - Medical Facility, Sheffield, Alabama
  - Medical Facility, Peoria, Arizona
  - Medical Facility3, Phoenix, Arizona
  - Medical Facility, Phoenix, Arizona
  - Medical Facility2, Phoenix, Arizona
  - Medical Facility, Tucson, Arizona
  - Medical Facility2, Hot Springs, Arkansas
  - Medical Facility, Hot Springs, Arkansas
  - Medical Facility, Bakersfield, California
  - Medical Facility, Chula Vista, California
  - Medical Facility, Fullerton, California
  - Medical Facility, Garden Grove, California
  - Medical Facility, Huntington Beach, California
  - Medical Facility 2, Huntington Park, California
  - Medical Facility, Huntington Park, California
  - Medical Facility, Irvine, California
  - Medical Facility, La Mesa, California
  - Medical Facility, Lancaster, California
  - Medical Facility, Lomita, California
  - Medical Facility2, Los Angeles, California
  - Medical Facility, Los Angeles, California
  - Medical Facility, Pomona, California
  - Medical Facility, Sacramento, California
  - Medical Facility, San Diego, California
  - Medical Facility, Upland, California
  - Medical Facility, Victorville, California
  - Medical Facility, Grand Junction, Colorado
  - Medical Facility, Lakewood, Colorado
  - Medical Facility, Aventura, Florida
  - Medical Facility, Boynton Beach, Florida
  - Medical Facility, Cape Coral, Florida
  - Medical Facility, Doral, Florida
  - Medical Facility, Edgewater, Florida
  - Medical Facility, Hialeah, Florida
  - Medical Facility, Hollywood, Florida
  - Medical Facility, Homestead, Florida
  - Medical Facility, Lake Worth, Florida
  - Medical Facility2, Lake Worth, Florida
  - Medical Facility, Leesburg, Florida
  - Medical Facility3, Miami, Florida
  - Medical Facility2, Miami, Florida
  - Medical Facility, Miami, Florida
  - Medical Facility9, Miami, Florida
  - Medical Facility5, Miami, Florida
  - Medical Facility8, Miami, Florida
  - Medical Facility6, Miami, Florida
  - Medical Facility7, Miami, Florida
  - Medical Facility4, Miami, Florida
  - Medical Facility, Miami Beach, Florida
  - Medical Facility, Miami Gardens, Florida
  - Medical Facility2, Miami Lakes, Florida
  - Medical Facility, Miami Lakes, Florida
  - Medical Facility, Orlando, Florida
  - Medical Facility2, Orlando, Florida
  - Medical Facility, Ormond Beach, Florida
  - Medical Facility, Pompano Beach, Florida
  - Medical Facility, Sweetwater, Florida
  - Medical Facility, Tamarac, Florida
  - Medical Facility, Tampa, Florida
  - Medical Facility3, Tampa, Florida
  - Medical Facility4, Tampa, Florida
  - Medical Facility2, Tampa, Florida
  - Medical Facility5, Tampa, Florida
  - Medical Facility, Winter Haven, Florida
  - Medical Facility3, Atlanta, Georgia
  - Medical Facility2, Atlanta, Georgia
  - Medical Facility, Atlanta, Georgia
  - Medical Facility, Decatur, Georgia
  - Medical Facility, Lawrenceville, Georgia
  - Medical Facility, Union City, Georgia
  - Medical Facility, Woodstock, Georgia
  - Medical Facility, Blackfoot, Idaho
  - Medical Facility2, Idaho Falls, Idaho
  - Medical Facility, Idaho Falls, Idaho
  - Medical Facility, Chicago, Illinois
  - Medical Facility, Eunice, Louisiana
  - Medical Facility, Mandeville, Louisiana
  - Medical Facility, Marrero, Louisiana
  - Medical Facility, Metairie, Louisiana
  - Medical Facility, New Orleans, Louisiana
  - Medical Facility2, New Orleans, Louisiana
  - Medical Facility, Prairieville, Louisiana
  - Medical Facility, Shreveport, Louisiana
  - Medical Facility, Columbia, Maryland
  - Medical Facility, Oxon Hill, Maryland
  - Medical Facility, Towson, Maryland
  - Medical Facility, Fayette, Mississippi
  - Medical Facility, Gulfport, Mississippi
  - Medical Facility, Jackson, Mississippi
  - Medical Facility, Ridgeland, Mississippi
  - Medical Facility, Great Falls, Montana
  - Medical Facility, Kalispell, Montana
  - Medical Facility, Missoula, Montana
  - Medical Facility2, Las Vegas, Nevada
  - Medical Facility, Las Vegas, Nevada
  - Medical Facility2, Albuquerque, New Mexico
  - Medical Facility, Albuquerque, New Mexico
  - Medical Facility, Brooklyn, New York
  - Medical Facility2, Brooklyn, New York
  - Medical Facility, Garden City, New York
  - Medical Facility, Schenectady, New York
  - Medical Facility, The Bronx, New York
  - Medical Facility, Charlotte, North Carolina
  - Medical Facility, Greensboro, North Carolina
  - Medical Facility, New Bern, North Carolina
  - Medical Facility, Winston-Salem, North Carolina
  - Medical Facility, Cincinnati, Ohio
  - Medical Facility2, Columbus, Ohio
  - Medical Facility, Columbus, Ohio
  - Medical Facility, Dayton, Ohio
  - Medical Facility2, Dayton, Ohio
  - Medical Facility, Lima, Ohio
  - Medical Facility, Middleburg Heights, Ohio
  - Medical Facility, Tulsa, Oklahoma
  - Medical Facility, Eugene, Oregon
  - Medical Facility, Portland, Oregon
  - Medical Facility, Beaver, Pennsylvania
  - Medical Facility, Scottdale, Pennsylvania
  - Medical Facility, Smithfield, Pennsylvania
  - Medical Facility, Upper Saint Clair, Pennsylvania
  - Medical Facility, Charleston, South Carolina
  - Medical Facility, Easley, South Carolina
  - Medical Facility, Greenville, South Carolina
  - Medical Facility, Lancaster, South Carolina
  - Medical Facility, Myrtle Beach, South Carolina
  - Medical Facility, Powdersville, South Carolina
  - Medical Facility, Seneca, South Carolina
  - Medical Facility, Summerville, South Carolina
  - Medical Facility2, Chattanooga, Tennessee
  - Medical Facility, Chattanooga, Tennessee
  - Medical Facility, Hendersonville, Tennessee
  - Medical Facility, Memphis, Tennessee
  - Medical Facility, Nashville, Tennessee
  - Medical Facility, Austin, Texas
  - Medical Facility, Carrollton, Texas
  - Medical Facility2, Carrollton, Texas
  - Medical Facility, Corpus Christi, Texas
  - Medical Facility, Dallas, Texas
  - Medical Facility, Frisco, Texas
  - Medical Facility, Georgetown, Texas
  - Medical Facility2, Houston, Texas
  - Medical Facility, Houston, Texas
  - Medical Facility, Kingwood, Texas
  - Medical Facility, League City, Texas
  - Medical Facility2, McKinney, Texas
  - Medical Facility, McKinney, Texas
  - Medical Facility2, Mesquite, Texas
  - Medical Facility, Mesquite, Texas
  - Medical Facility, Missouri City, Texas
  - Medical Facility, Pearland, Texas
  - Medical Facility2, Plano, Texas
  - Medical Facility, Plano, Texas
  - Medical Facility, San Antonio, Texas
  - Medical Facility 2, Sugar Land, Texas
  - Medical Facility3, Sugar Land, Texas
  - Medical Facility, Sugar Land, Texas
  - Medical Facility 2, Draper, Utah
  - Medical Facility, Draper, Utah
  - Medical Facility, Pleasant Grove, Utah
  - Medical Facility, Salt Lake City, Utah
  - Medical Facility, Falls Church, Virginia
  - Medical Facility, Manassas, Virginia
  - Medical Facility, Norfolk, Virginia
  - Medical Facility, Kingwood, West Virginia
  - Medical Facility, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Puttagunta S, Aronin SI, Gupta J, Das AF, Gupta K, Dunne MW. Sulopenem versus Amoxicillin/Clavulanate for the Treatment of Uncomplicated Urinary Tract Infection. NEJM Evid. 2025 Jul;4(7):EVIDoa2400414. doi: 10.1056/EVIDoa2400414. Epub 2025 Jun 24. PMID 40552968

RESULTS

PARTICIPANT FLOW:
Groups:
- Amoxicillin/Clavulanate: Amoxicillin/clavulanate 875 mg/125 mg PO twice daily for 5 days
  Amoxicillin/clavulanate: Oral Augmentin twice daily for 5 days
Period: Overall Study
Arm/Group | Sulopenem Etzadroxil/Probenecid | Amoxicillin/Clavulanate
Started | 1111 | 1111
Completed | 1057 | 1063
Not Completed | 54 | 48

BASELINE CHARACTERISTICS:
Population: Microbiological modified intent-to-treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Sulopenem Etzadroxil/Probenecid | Amoxicillin/Clavulanate | Total
Number analyzed (Participants) | 522 | 468 | 990
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (17.31) | 48.6 (17.18) | 49.5 (17.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 522 | 468 | 990
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 333 | 296 | 629
  Not Hispanic or Latino | 189 | 171 | 360
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 10 | 8 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 84 | 84 | 168
  White | 419 | 370 | 789
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 4 | 12
Region of Enrollment [Number; unit: participants] — Patients enrolled in the United States
  participants
    United States | 522 | 468 | 990
Diabetes [Count of Participants; unit: Participants] | 86 | 68 | 154

OUTCOME MEASURES:

1. Primary Outcome: Overall Success
Description: Clinical Success (resolution of uncomplicated urinary tract infection (uUTI) symptoms present at study entry and no new symptoms) AND Microbiologic success (eradication of the baseline pathogen)
Time Frame: Day 12+/-1 day
Population: Microbiologic Modified Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Sulopenem Etzadroxil/Probenecid | Amoxicillin/Clavulanate
Number analyzed (Participants) | 522 | 468
Participants | 318 | 260

2. Primary Outcome: Overall Success Susceptible Population
Description: as for outcome 1
Time Frame: Day 12+/-1 day
Population: Microbiological Modified intent-to-treat Susceptible Population
Measure: Count of Participants; unit: Participants
Arm/Group | Sulopenem Etzadroxil/Probenecid | Amoxicillin/Clavulanate
Number analyzed (Participants) | 480 | 442
Participants | 296 | 243

3. Secondary Outcome: Clinical Success Modified Intent-to-treat Population
Description: Resolution of uncomplicated urinary tract infection (uUTI) symptoms present at study entry and no new symptoms
Time Frame: Day 12+/-1 day
Population: Modified Intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Sulopenem Etzadroxil/Probenecid | Amoxicillin/Clavulanate
Number analyzed (Participants) | 1107 | 1107
Participants | 851 | 849

4. Secondary Outcome: Clinical Success
Description: Resolution of uncomplicated urinary tract infection (uUTI) symptoms present at study entry and no new symptoms
Time Frame: Day 12+/-1 day
Population: Microbiological Modified Intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Sulopenem Etzadroxil/Probenecid | Amoxicillin/Clavulanate
Number analyzed (Participants) | 522 | 468
Participants | 397 | 358

5. Secondary Outcome: Clinical Success Susceptible Population
Description: Resolution of uncomplicated urinary tract infection (uUTI) symptoms present at study entry and no new symptoms
Time Frame: Day 12+/-1 day
Population: Microbiological Modified Intent-to-treat Susceptible Population
Measure: Count of Participants; unit: Participants
Arm/Group | Sulopenem Etzadroxil/Probenecid | Amoxicillin/Clavulanate
Number analyzed (Participants) | 480 | 442
Participants | 371 | 339

6. Secondary Outcome: Microbiologic Success
Description: Eradication of the Baseline Pathogen
Time Frame: Day 12+/-1 day
Population: Microbiological Modified Intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Sulopenem Etzadroxil/Probenecid | Amoxicillin/Clavulanate
Number analyzed (Participants) | 522 | 468
Participants | 390 | 315

7. Secondary Outcome: Microbiologic Success Susceptible Population
Description: Microbiologic Success: Eradication of the Baseline Pathogen
Time Frame: Day 12+/-1 day
Population: Microbiological Modified Intent-to-treat Susceptible Population
Measure: Count of Participants; unit: Participants
Arm/Group | Sulopenem Etzadroxil/Probenecid | Amoxicillin/Clavulanate
Number analyzed (Participants) | 480 | 442
Participants | 361 | 295

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Sulopenem Etzadroxil/Probenecid | Amoxicillin/Clavulanate
All-Cause Mortality (participants affected / at risk) | 0/1107 | 0/1107
Serious Adverse Events (participants affected / at risk) | 0/1107 | 5/1107
Other Adverse Events (participants affected / at risk) | 198/1107 | 118/1107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sulopenem Etzadroxil/Probenecid (N=1107) | Amoxicillin/Clavulanate (N=1107)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sulopenem Etzadroxil/Probenecid (N=1107) | Amoxicillin/Clavulanate (N=1107)
Diarrhea (Gastrointestinal disorders) | 90 (90) | 45 (45) — Treatment-emergent Diarrhea
Nausea (Gastrointestinal disorders) | 48 (48) | 48 (48) — Treatment-emergent nausea
Headache (Nervous system disorders) | 24 (24) | 17 (17) — Treatment-emergent Headache
Vulvovaginal mycotic infection (Infections and infestations) | 20 (20) | 4 (4) — Treatment-emergent Vulvovaginal mycotic infection
Vomiting (Gastrointestinal disorders) | 16 (16) | 4 (4) — Treatment-emergent Vomiting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT05584657/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT05584657/SAP_001.pdf